CLINICAL TRIAL: NCT06675318
Title: The Effect of Contralateral Isokinetic Lower Extremity Exercises Added to Conventional Rehabilitation in Unilateral Painful Knee Osteoarthritis
Brief Title: The Effect of Contralateral Isokinetic Lower Extremity Exercises in Unilateral Painful Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Emine METIN IPEK, Research Assistant, Physical Medicine and Rehabilitation, Principal Investigator, M.D., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Contralateral Exercise
Record Dates: First submitted 2024-07-13; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Exercise
Keywords: Knee osteoarthritis; Isokinetic exercise; Contralateral exercise effect; Quadriceps muscle thickness; Physical Function; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: A prospective cohort study involving two parallel groups with randomization control
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical and demographic data collection and statistical analyses will be conducted by a blinded researcher with respect to the treatment group and clinical findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients with unilateral painful knee osteoarthritis who are applied to Gazi University Faculty of Medicine PM&R will be included. 20 sessions of conventional physical therapy and rehabilitation (isometric exercises, TENS, hot pack) for the symptomatic extremity will be applied to patients In the active control group.
  Interventions: Other: Quadriceps isometric exercises, along with hot pack and TENS for painful knee
- Study group (Experimental): Patients with unilateral painful knee osteoarthritis who are applied to Gazi University Faculty of Medicine PM&R will be included. 20 sessions of conventional physical therapy and rehabilitation for the symptomatic extremity combined with isokinetic strengthening exercises for the asymptomatic extremity will be applied to patients In the experimental group
  Interventions: Other: Cross training for quadriceps muscle of contralateral lower limb; Other: Quadriceps isometric exercises, along with hot pack and TENS for painful knee

INTERVENTIONS:
Other: Cross training for quadriceps muscle of contralateral lower limb — An isokinetic exercise program consisting of 20 sessions conducted five days a week. The program begins with five repetitions at a speed of 60°/s, followed by sets of 5-15 repetitions with incremental increases of 30°/s. Rest periods of 30 seconds were included between sets.
  Arms: Study group
Other: Quadriceps isometric exercises, along with hot pack and TENS for painful knee — 10 repetitions of quadriceps isometric exercises in 3 sets, along with hot pack and TENS treatments for painful knee

SUMMARY:
Patients with unilateral knee pain due to knee osteoarthritis presenting to our clinic will be included in a 20-session treatment program, either on an outpatient basis or as inpatients at our clinic. The patients will be divided into 2 groups, and conventional treatments including isometric exercises, TENS (Transcutaneous Electrical Nerve Stimulation) and hot pack therapy for the painful knee will be administered to both groups. In addition to these treatments, the intervention group will receive isokinetic exercise sessions using the Cybex 770 Norm isokinetic dynamometer system (Lumex Inc., Ronkonkoma, New York) at speeds of 60°/s and 180°/s according to the device's standard protocol, targeting the contralateral lower extremity. Subsequently, examinations and measurements will be conducted to evaluate patients for reduction in pain, increase in muscle strength, improvement in functionality, and increase in thigh muscle thickness.

DETAILED DESCRIPTION:
Osteoartritis is the most common form of arthritis, originating from the failed repair of joint damage caused by stress initiated by any joint or periarticular tissue abnormality. Its most common symptom is pain. The long-term consequences of osteoarthritis include decreased physical activity, loss of conditioning, sleep disturbances, fatigue, depression, and disability. Factors associated with increased risk of knee osteoarthritis include advanced age, female gender, overweight or obesity, knee injury, occupational factors, and varus or valgus alignment of the knee.

With the increasing aging population, degenerative joint problems have become relevant to a large portion of society. Exercise is a fundamental component in the treatment of this chronic disease, which limits functionality and reduces quality of life.

A systematic review including 32 randomized controlled trials evaluating 5362 participants showed that various types of exercise provide improvement in pain, functionality, and quality of life in knee osteoarthritis.

Musculoskeletal pains can lead to cortical reorganization in both somatosensory and motor areas, which can reduce motor activity in both the affected and unaffected contralateral extremities. For example, a decrease in motor activity in both painful and pain-free contralateral extremities has been identified during acute pain and/or in the presence of chronic pain.

If exercise is performed to increase muscle strength on one side of the body, strength may also increase on the opposite side. This effect, called the contralateral exercise phenomenon, is typically measured in homologous muscles. Although known for over a century, most studies have not been well-designed to demonstrate the exact magnitude of the strength increase effect. However, an updated meta-analysis of 16 studies indicates that the size of the contralateral exercise effect is approximately 8% of baseline strength or about half of the increase in strength on the exercised side.

However, there are few studies examining the combined effects of contralateral lower extremity isokinetic exercises on pain, muscle thickness, and functionality. Therefore, the aim of this study is to demonstrate the effect of isokinetic exercises applied to the contralateral lower extremity added to routine treatment on muscle strength, muscle thickness, and functionality in the painful knee, and to show its potential relationship. We aim to provide clinicians with a new perspective on the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study
* To be aged 50 years or older
* To have a clinically and radiographically confirmed diagnosis of knee osteoarthritis
* To have unilateral knee pain due to osteoarthritis (VAS <2 in the contralateral knee, VAS >2 in the painful knee)
* To have Kellgren-Lawrence Grade 1-3 in the painful knee and Kellgren-Lawrence Grade <4 in the contralateral knee
* To have dominance of the right lower extremity

Exclusion Criteria:

* A history of previous lower extremity fractures or orthopedic surgery that would interfere with isokinetic and isometric exercises in both lower extremities
* The presence of significant sensorimotor deficits due to neurological diseases
* The presence of known inflammatory rheumatic diseases
* The presence of non-curable malignant tumors with bone metastasis
* The presence of neuropsychiatric diseases or conditions that would hinder cooperation
* Having undergone interventions such as injections for pain relief within the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) score | From enrollment day to the end of the rehabilitation program at 4 weeks.
  WOMAC score evaluation following the last treatment session. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, validated questionnaire designed to assess pain, stiffness, and physical function in patients with knee and hip osteoarthritis. It consists of 24 items divided into three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Patients rate their symptoms on a Likert scale, with higher scores indicating worse pain, stiffness, or functional limitations. The WOMAC is commonly used in clinical research to evaluate the efficacy of various treatments for osteoarthritis.

SECONDARY OUTCOMES:
Pain level; VAS score | From enrollment day to the end of the rehabilitation program at 4 weeks
  The Visual Analog Scale (VAS) is a tool used to measure a patient's level of pain. It consists of a straight line with endpoints defining extreme limits such as 'no pain' and 'worst pain imaginable.' The patient marks on the line the point that they feel represents their perception of their current state. This method is simple, reliable, and widely used in both clinical and research settings to quantify pain intensity.
Muscle strength | From enrollment day to the end of the rehabilitation program at 4 weeks
  To evaluate isokinetic muscle strength, the Cybex 770 Norm isokinetic dynamometer system (Lumex Inc., Ronkonkoma, New York) will be used to measure peak torque values for flexion and extension at a speed of 60°/s, peak torque values for flexion and extension at a speed of 180°/s, and total work production (endurance) at 180 degrees.
Physical function | From enrollment day to the end of the rehabilitation program at 4 weeks
  To evaluate physical function, SF-36 (Short Form-36) will be used. SF-36: The SF-36 is a scale consisting of 36 items divided into 8 subscales: physical functioning, physical role, emotional role, pain, general health, energy, social functioning, and mental health. Lower scores indicate higher levels of restriction. The Turkish version has been validated for reliability and validity.
Lower extremity function | From enrollment day to the end of the rehabilitation program at 4 weeks
  To evaluate physical function, TUG test will be used. Timed Up and Go Test (TUG): To assess lower extremity function, participants will be timed as they rise from a chair, walk to a marked point 3 meters away, turn around, and return to sit in the chair. The elapsed time will be recorded.
Ultrasonographic Measurement of Thigh muscle thickness | From enrollment day to the end of the rehabilitation program at 4 weeks
  Participants will be evaluated in a supine position. Measurements will be taken for the Rectus Femoris (RF), Vastus Intermedius (VI), Vastus Lateralis (VL), Vastus Medialis (VM), and Vastus Medialis Obliquus (VMO) muscles. A line will be drawn from the upper pole of the patella to the anterior superior iliac spine (ASIS) along the length of the thigh. RF and VI will be measured at 50% of this line. For VL, the circumference of the thigh at 50% of the line will be measured, and then VL will be measured at 10% of the circumference. VM will be measured at 20% of the line, and then at 12.5% of the circumference at the same point. VMO will be measured 4 cm above and 3 cm medial to the upper pole of the patella.
  MyLab 70 XV ultrasound device (Esaote Biomedica, Genoa, Italy) with a multifrequency linear probe will be used at the Physical Medicine and Rehabilitation Unit of Gazi University Faculty of Medicine.
Range of motion | From enrollment day to the end of the rehabilitation program at 4 weeks
  Range of motion will be measured with a goniometer according to the neutral zero method.
  The principle of joint measurement by the neutral zero method is to measure the movement of a joint from a defined neutral O-position. The measured angle gives the magnitude of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Jale Meray, MD, Study Director — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Hawker GA, Stewart L, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Gooberman-Hill R. Understanding the pain experience in hip and knee osteoarthritis--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):415-22. doi: 10.1016/j.joca.2007.12.017. Epub 2008 Mar 4. PMID 18296075
- [Background] Flor H. Cortical reorganisation and chronic pain: implications for rehabilitation. J Rehabil Med. 2003 May;(41 Suppl):66-72. doi: 10.1080/16501960310010179. PMID 12817660
- [Background] Arguis MJ, Perez J, Martinez G, Ubre M, Gomar C. Contralateral neuropathic pain following a surgical model of unilateral nerve injury in rats. Reg Anesth Pain Med. 2008 May-Jun;33(3):211-6. doi: 10.1016/j.rapm.2007.12.003. PMID 18433671
- [Background] Cheon S, Lee JH, Jun HP, An YW, Chang E. Acute Effects of Open Kinetic Chain Exercise Versus Those of Closed Kinetic Chain Exercise on Quadriceps Muscle Thickness in Healthy Adults. Int J Environ Res Public Health. 2020 Jun 29;17(13):4669. doi: 10.3390/ijerph17134669. PMID 32610511
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067